CLINICAL TRIAL: NCT04648189
Title: Are Anti-EGFR Monoclonal Antibodies the Magic Bullets That Remove Circulating EGFR+EpCAM+ Tumor Cells in Patients With Non-small Cell Lung Cancer
Brief Title: Cetuxibab to Reduce Circulating Tumor Cells in Early Stage NSCLC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: One of the participating specialties has decided to no longer cooperate in this research
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M20EGF
Record Dates: First submitted 2020-11-13; First posted 2020-12-01 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Lung Cancer; Surgery; Circulating Tumor Cell
MeSH Terms: conditions — Lung Neoplasms; Neoplastic Cells, Circulating | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single dose cetuximab prior to surgery (Experimental): A single dose of cetuximab, 400mg/m2, will be administered 72 to 48 hours prior to surgery
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — A single dose of cetuximab, 400mg/m2, will be administered 72 to 48 hours prior to surgery

SUMMARY:
Cetuximab to reduce the amound of circulating tumor cells in early stage NSCLC

DETAILED DESCRIPTION:
A multicenter single arm phase II trial. 40 patients with pathology proven stage I-IIIA NSCLC that are eligible for resection will be enrolled in this study. All patients will receive one dose of cetuximab prior to surgery. Blood will be drawn on multiple timepoints to assess te amount of circulating tumor cells

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Presence of surgically resectable NSCLC, stage I-IIIA, with curative intent surgery planned.
* ≥10 EGFR+EpCAM+ cells detected in the baseline blood sample.
* Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must agree to use adequate barrier birth control measures (e.g., cervical cap, condom, and diaphragm) during the course of the trial. Oral birth control methods alone will not be considered adequate on this study, because of the potential pharmacokinetic interaction between study drug and oral contraceptives. Concomitant use of oral and barrier contraceptives is advised. Contraception is necessary for at least 6 months after receiving study drug

Exclusion Criteria:

* Chemotherapy or other anti-cancer therapy including radiotherapy during the study or within 4 weeks prior to the start of the study.
* Prior anti-EGFR mAb therapy
* Other currently active malignancy
* Immunosuppressive drugs during the study or within 4 weeks prior to the start of te study
* Expected adverse reactions/allergies or study medication
* Mental disorder/unable to give informed consent
* Pregnancy or breast-feeding patients
* Significant skin condition interfering with treatment
* Major surgery within 28 days before start of study.
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results.
* Any condition that is unstable or could jeopardize the safety of the subject and their compliance in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
reduction of circulating tumor cells | From date of registration until CTC measurement at 3 months after surgery.
  The primary objective of this study is to determine whether a single neoadjuvant dose of cetuximab (anti-EGFR mAb) - administered 72 to 48 hours prior to surgery - will reduce the number of CTCs in patients. The reduction of CTCs will be expressed in percentage as more or less than 50% changed from baseline.

SECONDARY OUTCOMES:
the reduction of CTC's in percentage as a continuous variable | From date of registration until CTC measurement at 3 months after surgery.
  the reduction of CTC's in percentage as a continuous variable will be assesed
plasma ability killing tumor cells | From date of registration until CTC measurement at 3 months after surgery.
  the concentration of plasma who have the ability to inhibit growth in patients treated with cetuximab, ADCP and/or ADCC of tumor cells by cytotoxic immune effector cells
disease free survival | From date of surgery to until the date of first documented progression or date of death from any cause.
  Although this study is not powered for disease free survival, we will conduct follow-up of all the patients in order to get preliminary information about potential clinical efficacy
safety | From date of registration until CTC measurement at 3 months after surgery.
  Safety and toxicity will also be studied. All adverse events and SUSARS will be scored using the common Terminology Criteria for Adverse Events (CTCAE).

CONTACTS AND LOCATIONS:
Overall Officials: Egbert Smit, prof, Principal Investigator — The Netherlands Cancer Institute-Antoni van Leeuwenhoek; Marjolein van Egmond, prof, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (2):
- Netherlands (2):
  - Amsterdam UMC - VUMC, Amsterdam
  - Leiden University Medical Center, Leiden

IPD SHARING:
Plan to Share IPD: Undecided
to be decided